CLINICAL TRIAL: NCT04715087
Title: Staphylococcus Aureus in Atopic Dermatitis Immunopathology
Acronym: STADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL18_0732; 2020-A01547-32 (Other: ID-RCB)
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Staphyloccocus aureus; Immunopathology
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atopic dermatitis patients (Other): Bacteriological skin swab samples from AD patients will be performed at screening visit. Each sample will be cultured and isolated to be re-applied (via patchtest) to AD patient. After reading the patch test results, skin biopsies will be performed
  Interventions: Other: Blood sample (Day -42 to Day -28, Day 3),Skin swab sampling (Day -42 to Day -28, Day 0, Day 13) , patch test application (Day 0) , skin biopsies (Day 13)
- Healthy controls (Other): Bacteriological skin swab samples from AD patients will be performed at screening visit. Each sample will be cultured and isolated to be applied (via patchtest) to a paired (age/sex) healthy volunteer. After reading the patch test results, skin biopsies will be performed.
  Interventions: Other: Blood sample (Day 0 ,Day 3),Skin swab sampling (Day 0,Day 13), patch test application (Day 1), skin biopsies (Day 13)

INTERVENTIONS:
Other: Blood sample (Day -42 to Day -28, Day 3),Skin swab sampling (Day -42 to Day -28, Day 0, Day 13) , patch test application (Day 0) , skin biopsies (Day 13) — A 50 mL blood sample will be collected in Lithium Heparin tubes (45 mL) and dry tube (5 mL), by venipuncture, at screening and Day 3. Bacteriological samples from AD patients will be performed by swabbing the skin at screening visit (Day -42 to Day -28). Each sample will be cultured in a RPMI/human serum AB medium and methi.R (methicillin Resistant) strains will be eliminated. Thus, only S. aureus methi.S (methicillin Sensitive) will be isolated to be re-applied (via patchtest) to AD patient. A well-characterized S. epidermidis lab strain will be also applied to AD patients. Patch tests containing S. aureus, S. epidermidis or a mix S. aureus/S. epidermidis will be applied on healed or improved area as defined by a lesional score ≤ 1 or a 2-point change from the baseline lesional score. Patch tests will be applied 48h and reading of the patch tests results and biopsies will be performed 72h after patch test application.
  Arms: Atopic dermatitis patients
Other: Blood sample (Day 0 ,Day 3),Skin swab sampling (Day 0,Day 13), patch test application (Day 1), skin biopsies (Day 13) — A 50 mL blood sample will be collected in Lithium Heparin tubes (45 mL) and dry tube (5 mL), by venipuncture, at Day 0 and Day 3.
  Each bacteriological sample from AD patients performed by swabbing the skin at screening visit will be cultured in a RPMI/human serum AB medium and methi.R (methicillin Resistant) strains will be eliminated. Thus, only S. aureus methi.S (methicillin Sensitive) will be isolated to be applied (via patchtest) to a paired (age/sex) healthy volunteer. A well-characterized S. epidermidis lab strain will be also applied to healthy volunteers. Patch tests containing S. aureus, S. epidermidis or a mix S. aureus/S. epidermidis will be applied on healthy skin. Patch tests will be applied 48h and reading of the patch tests results and biopsies will be performed 72h after patch test application
  Arms: Healthy controls

SUMMARY:
Atopic Dermatitis (AD) is a frequent inflammatory skin disease characterized by recurrent eczema. It associates genetic/epigenetic-induced alterations of epidermal barrier and type-2 inflammation/hypersensitivity, which may be triggered by different antigens that pass through the altered skin . Some studies have reported that environmental pathogens such as house dust mites are able to induce type-2 inflammation through particular activation of innate immunity .

Multiple staphylococcal strains are commonly found on the skin of AD patients. Interestingly, recent findings suggest that S. aureus may be a key factor of AD inflammation: (i) 90% of AD patients have S. aureus skin colonization on lesional skin , (ii) AD patients with S. aureus skin colonization have more increased type-2 inflammatory markers in comparison with AD patients without SA skin colonization , (iii) skin colonization by monoclonal S. aureus strains correlate with severe flares and (iv) S. aureus is detected in both epidermis and dermis during AD flares; In this study, our hypothesis is that S. aureus induces AD flares through a type 2 T cell-mediated hypersensitivity against S. aureus, involving innate and adaptive responses. Conversely, S. epidermidis, a commensal strain, has a protective effect against S. aureus dysbiosis. To this end, we will characterize, in the skin and the blood, the immune response induced by cutaneous application of : i) S. aureus isolated from patients with moderate-to-severe AD which will mimic the cutaneous dysbiosis occurring in the natural course of AD; ii) S. aureus toxins without bacteria to evaluate the skin response against those particular proteins; iii) a laboratory strain of S. epidermidis, a common well-tolerated skin commensal bacteria; iv) a mix of S. aureus and S. epidermidis to evaluate the regulatory effect of S. epidermidis on the S. aureus-induced AD inflammation.

Importantly, this characterization will be led in AD patients (with alterations of skin barrier), compared to healthy volunteers (without alterations of skin barrier), as controls.

ELIGIBILITY:
Inclusion Criteria:

* Subject over 18 years of age
* Subject able to read, understand and give documented informed consent
* Subject who gave written informed consent
* Subject willing and able to comply with the protocol requirements for the duration of the study
* Subjects with health insurance coverage according to local regulations
* For woman with childbearing potential;

  * Use of a highly effective method of birth control from at least 1 month prior to study enrollment until the last visit
  * Negative urine pregnancy test at inclusion visit
* Subject with I, II, III or IV skin phototype (according to Fitzpatrick scale)
* Subject accepting patch-tests and skin biopsies Specific criteria for AD patients
* Subject diagnosed with moderate-to-severe AD, defined as EASI ≥7 and DLQI ≥ 6
* Subject with AD involvement of ≥ 5% of Body Surface Area (BSA)
* Subject with at least one AD lesion:

  * Located either on upper extremities (except hands) or lower extremities (except feet)
  * With a sufficient extent to allow all the investigations
  * With a lesional area score ≥ 6

Exclusion Criteria:

* Pregnancy or breast-feeding women, or planning to become pregnant or breastfeed during the study
* History of allergic reaction to local anesthetic product
* History of wound healing disorders (e.g. hypertrophic scars, keloids)
* Subject with known active infection to HBV, HCV or HIV
* Subject with known blood dyscrasia
* Subject having applied topical immunomodulators, non-steroidal anti-inflammatory, corticoids, antihistamines, antibiotics or disinfectants on investigational limbs within 1 week before the inclusion visit
* Subject treated with cyclosporine, methotrexate oral corticosteroids, azathioprine, mycophenolate-mofetil, and/or any other systemic immunosuppressor/immunomodulator within 4 weeks before the study
* Subject treated by a biologic therapy within 3 months before the study
* Subject treated with ultraviolet therapy within 4 weeks before study
* Subject presenting clinically significant medical disease that is uncontrolled despite treatment that is likely, in the opinion of the investigator, to impact patient's ability to participate in the study or to impact the study efficacy or safety assessments
* Subject treated with an investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer, before the baseline visit
* Subject with immunocompromised people in its close circle
* Subject protect by the law (adult under guardianship, or hospitalized in a public or private institution for a reason other than study, or incarcerated)
* Subject in an exclusion period from a previous study or who is participating in another clinical trial
* Specific criteria for AD patients :

  o Subject currently experiencing or having a history of other concomitant skin conditions that would interfere with evaluation of AD
* Specific criteria for healthy control :

  * Subject currently experiencing or having an history of AD or other concomitant condition that would interfere with evaluation of skin reaction induced by patch test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of a clinical inflammatory skin lesion after application of patch test containing a solution of methi-sensible (methi-S) S.aureus, in AD patients or healthy volunteers. | Day 3
  A difference of the local AD severity will be searched between baseline and after S. aureus patch test application (in AD patients and healthy volunteers) according to the lesional scoring and the patch test scoring. A logistic mixed effects model will be performed to model the occurrence of clinical inflammatory skin lesion. For each sub-population (AD patients or healthy volunteers), a linear mixed effect model will be used to model the lesional scoring.

SECONDARY OUTCOMES:
Molecular analysis of cytokine skin expression induced by S.aureus patch test. | Day 3
  Results will be expressed as fold change compared to control skin from the same individual (qPCR analysis).
  * Type 2 inflammation: interleukins (IL)-4, 5, 13, 31
  * Type 1 inflammation: TNF, IFNγ
  * Type 17-22 inflammation: IL-12, IL-23, IL-17a, IL-22
  * Innate inflammation: TSLP, IL-25, IL-33, IL-1b, IL-1a, IL-18
  Then, a significant difference of each parameter cited above will also be searched between baseline and after S. aureus patch test application (in AD patients and healthy volunteers).
Type 2 specific cellular and molecular regulatory and inflammatory response in blood - OPTIONAL (only in case of additional funding/grant) | Day 3
  A significant difference of parameters will be searched between baseline and after S. aureus patch test application (in AD patients and healthy volunteers)
Presence/identification of S. aureus-specific virulence factors inducing a sensitization (immunoblotting) - OPTIONAL (only in case of additional funding/grant) | Day 3
  A significant difference of parameters will be searched between baseline and after S. aureus patch test application (in AD patients and healthy volunteers).
Differences in clinical skin response against S. epidermidis and mix S. aureus/S. epidermidis. | Day 3
  Results will be expressed as fold change compared to control skin from the same individual (qPCR analysis).
  * Type 2 inflammation: interleukins (IL)-4, 5, 13, 31)
  * Type 1 inflammation: TNF, IFNγ
  * Type 17-22 inflammation: IL-12, IL-23, IL-17a, IL-22
  * Innate inflammation: TSLP, IL-25, IL-33, IL-1b, IL-1a, IL-18
  Then, a significant difference of each parameter cited above will also be searched between S. epidermidis alone, mix S. epidermidis/S. aureus and S. aureus alone patch tests.
Molecular analysis of cytokine skin expression induced by S. epidermidis and mix S. aureus/S. epidermidis. | Day 3
  Results will be expressed as fold change compared to control skin from the same individual (qPCR analysis).
  * Type 2 inflammation: interleukins (IL)-4, 5, 13, 31)
  * Type 1 inflammation: TNF, IFNγ
  * Type 17-22 inflammation: IL-12, IL-23, IL-17a, IL-22
  * Innate inflammation: TSLP, IL-25, IL-33, IL-1b, IL-1a, IL-18
  Then, a significant difference of each parameter cited above will also be searched between S. epidermidis alone, mix S. epidermidis/S. aureus and S. aureus alone patch tests. A linear mixed effects model will be used to model each parameter of the molecular analysis of cytokine skin expression.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey NOSBAUM, MD, PhD, Principal Investigator — Allergy and Clinical Immunology Department - Centre Hospitalier Lyon Sud
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No